CLINICAL TRIAL: NCT00690950
Title: Switch Study: Are There Any Measurable Differences When Switching Patients on Finasteride Therapy to Dutasteride?
Brief Title: A Study to Determine the Improvement of the Symptoms of Benign Prostatic Hyperplasia (BPH) When Switching Subjects From Proscar to Avodart
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Urologic Consultants of Southeastern PA (Other)
Responsible Party: Dr. Richard C. Harkaway, Urologic consultants of Southeastern PA
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110895
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: BPH
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dutasteride — 0.5mg capsule, taken once daily for 12 months

SUMMARY:
Hypothesis: Dutasteride will perform better than finasteride in decreasing prostate volume, improving symptoms based on International Prostate Symptom score,and lower pvr based on the scientific information that dutasteride inhibits both Type I and II 5-alpha-reducatase vs. finasteride which only inhibits the Type II enzyme

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 50-80
* On finasteride for no less than 12 months
* Willing to undergo all necessary test in the 12 month evaluation

Exclusion Criteria:

* History of medication non-compliance
* Unwillingness to undergo/tolerate 2 blood draws
* Unwillingness to tolerate/undergo 2 TRUSP

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Laboratory parameters: including serum testosterone, DHT level and PSA | 12 months

SECONDARY OUTCOMES:
volume measurements of TRUSP and PVR | 12 months
A decrease in the AUASI | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Urologic Consultants of Southeastern PA, Bala-Cynwyd, Pennsylvania, United States